CLINICAL TRIAL: NCT01179516
Title: A Phase 3, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Fixed-Dose Study Comparing the Efficacy and Safety of 2 Doses (10 and 15 mg) of Lu AA21004 in Acute Treatment of Adults With Major Depressive Disorder
Brief Title: Safety and Efficacy Study of Vortioxetine (Lu AA21004) in Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LuAA21004_317; U1111-1116-3223 (Registry Identifier: WHO); SU-06032011-7846 (Registry Identifier: SMCTD)
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-10

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder; Depression; Drug Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Vortioxetine placebo-matching capsules, orally, once daily for up to 8 weeks.
  Interventions: Drug: Placebo
- Vortioxetine 10 mg (Experimental): Vortioxetine 10 mg, encapsulated tablets, orally, once daily for up to 8 weeks.
  Interventions: Drug: Vortioxetine
- Vortioxetine 15 mg (Experimental): Vortioxetine 10 mg, encapsulated tablets, orally, once daily for one week, then vortioxetine 15 mg, encapsulated tablets, orally, once daily for up to 7 weeks.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Encapsulated vortioxetine immediate release tablets
  Other Names: Lu AA21004; Brintellix®
  Arms: Vortioxetine 10 mg; Vortioxetine 15 mg
Drug: Placebo — Vortioxetine placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of vortioxetine, once daily (QD), compared with placebo in adults with major depressive disorder.

DETAILED DESCRIPTION:
The drug that was tested in this study is called Vortioxetine. Vortioxetine is being tested to treat depression in adults who have major depressive disorder (MDD). This study looked at MDD relief in people who took varying dosages of vortioxetine.

The study enrolled 469 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the three treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there was an urgent medical need):

* Vortioxetine 10 mg
* Vortioxetine 15 mg
* Placebo (dummy inactive capsule) - this was a capsule that looked like the study drug but had no active ingredient.

All participants were asked to take one capsule at the same time each day throughout the study.

This multi-center trial was conducted in the United States. The overall time to participate in this study was up to 14 weeks. Participants made 7 visits to the clinic, and were contacted by telephone 4 weeks after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Suffers from a major depressive episode (MDE) recurrent as the primary diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria.
* The reported duration of the current MDE is at least 3 months.
* Has a Montgomery Åsberg Depression Rating Scale (MADRS) total score of 26 or greater at Screening and Baseline Visits.
* Has a Clinical Global Impression - Severity of Illness (CGI-S) score of 4 or greater at Screening and Baseline Visits.

Exclusion Criteria:

* Has received any investigational compound <30 days before Screening or 5 half-lives prior to Screening.
* Has received Lu AA21004 in a previous clinical study.
* Has 1 or more the following:

  1. Any current psychiatric disorder other than MDD as defined in the DSM-IV-TR .
  2. Current or history of: manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
  3. Diagnosis of alcohol or other substance abuse or dependence (excluding nicotine or caffeine) as defined in the DSM-IV-TR that had not been in sustained full remission for at least 2 years prior to Screening.
  4. Presence or history of a clinically significant neurological disorder (including epilepsy).
  5. Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc).
  6. Any Axis II disorder that might compromise the study.
* The current depressive symptoms of the patient were considered by the investigator to have been resistant to 2 adequate antidepressant treatments of at least 6 weeks duration each.
* Has received electroconvulsive therapy, vagal nerve stimulation, or repetitive transcranial magnetic stimulation within 6 months prior to Screening.
* Was currently receiving formal cognitive or behavioral therapy, systematic psychotherapy, or planned to initiate such therapy during the study.
* Has a significant risk of suicide according to the investigator's clinical judgment or had a score ≥5 on item 10 (suicidal thoughts) of the MADRS or had made a suicide attempt in the previous 6 months.
* Was required to take excluded medications or it was anticipated that would require treatment with at least 1 of the disallowed concomitant medications during the study.
* Has a clinically significant unstable illness, for example hepatic impairment or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, rheumatologic, immunologic, hematological, infectious, dermatological disorder or metabolic disturbance. NOTE: For the purposes of this study, the following conditions were considered unstable due to the potential impact on assessment of MDD response: pain disorder, chronic fatigue syndrome, fibromyalgia, and obstructive sleep apnea.
* Has 1 or more laboratory value outside the normal range, based on the blood or urine samples taken at the Screening Visit, that were considered by the investigator to be clinically significant; or the patient has any of the following values at the Screening Visit:

  1. A serum creatinine value >1.5 times the upper limits of normal (× ULN).
  2. A total serum total bilirubin value >1.5 × ULN.
  3. A serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >2 × ULN.
* Has a thyroid stimulating hormone value outside the normal range.
* Has clinically significant abnormal vital signs.
* Has an abnormal electrocardiogram.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (61):
- United States (61):
  - Little Rock, Arkansas
  - Carson, California
  - Cerritos, California
  - El Centro, California
  - Fresno, California
  - Glendale, California
  - Los Angeles, California
  - Oakland, California
  - Oceanside, California
  - San Diego, California
  - Santa Ana, California
  - Sherman Oaks, California
  - Stanford, California
  - Upland, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Hockessin, Delaware
  - Fort Walton Beach, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - Pompano Beach, Florida
  - Atlanta, Georgia
  - Hoffman Estates, Illinois
  - Naperville, Illinois
  - Oak Brook, Illinois
  - Indianapolis, Indiana
  - Lafayette, Indiana
  - Newburgh, Indiana
  - Prarie Ridge, Kansas
  - Wichita, Kansas
  - Baltimore, Maryland
  - Fall River, Massachusetts
  - Watertown, Massachusetts
  - Clinton Township, Michigan
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Nashua, New Hampshire
  - Albuquerque, New Mexico
  - Staten Island, New York
  - Avon Lake, Ohio
  - Beachwood, Ohio
  - Canton, Ohio
  - Garfield Heights, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Salem, Oregon
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Lincoln, Rhode Island
  - Columbia, South Carolina
  - Franklin, Tennessee
  - Dallas, Texas
  - DeSoto, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Salt Lake City, Utah
  - Roanoke, Virginia
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Mahableshwarkar AR, Jacobsen PL, Serenko M, Chen Y, Trivedi MH. A randomized, double-blind, placebo-controlled study of the efficacy and safety of 2 doses of vortioxetine in adults with major depressive disorder. J Clin Psychiatry. 2015 May;76(5):583-91. doi: 10.4088/JCP.14m09337. PMID 26035186

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 65 investigative sites in the United States from 11 August 2010 to 04 June 2012.
Pre-assignment Details: Participants with a diagnosis of major depressive disorder were enrolled equally in 1 of 3 treatment groups, once a day placebo, 10 mg, or 15 mg vortioxetine.
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 15 mg
Started | 160 | 157 | 152
Treated | 160 | 154 | 151
Completed | 133 | 131 | 121
Not Completed | 27 | 26 | 31
Not completed — Pretreatment Event or Adverse Event | 6 | 8 | 12
Not completed — Lack of Efficacy | 4 | 2 | 0
Not completed — Noncompliance with Study Drug | 2 | 0 | 1
Not completed — Protocol Deviations | 4 | 3 | 3
Not completed — Withdrawal of Consent | 2 | 6 | 10
Not completed — Lost to Follow-up | 7 | 7 | 3
Not completed — Other | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 15 mg | Total
Number analyzed (Participants) | 160 | 157 | 152 | 469
Age Continuous [Mean (Standard Deviation); unit: years] | 46.2 (11.79) | 45.2 (11.94) | 43.8 (13.51) | 45.1 (12.44)
Age, Customized [Number; unit: participants]
  ≤55 years | 122 | 129 | 120 | 371
  >55 years | 38 | 28 | 32 | 98
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 113 | 108 | 329
  Male | 52 | 44 | 44 | 140
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 20 | 16 | 18 | 54
  Non-Hispanic and non-Latino | 140 | 141 | 134 | 415
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (White, including Hispanic) | 124 | 115 | 109 | 348
  Black | 35 | 39 | 38 | 112
  Asian | 1 | 1 | 4 | 6
  American Indian or Alaska Native | 0 | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 160 | 157 | 152 | 469
Height [Mean (Standard Deviation); unit: cm] | 168.85 (10.407) | 167.35 (9.523) | 167.52 (9.789) | 167.92 (9.920)
Weight [Mean (Standard Deviation); unit: kg] | 89.14 (24.010) | 87.74 (23.914) | 86.49 (23.154) | 87.81 (23.678)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.14 (7.533) | 31.29 (8.063) | 30.78 (7.752) | 31.07 (7.771)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 99.93 (17.820) | 100.02 (16.762) | 97.93 (17.536) | 99.31 (17.370)
Smoking Classification [Number; unit: participants]
  Never smoked | 83 | 86 | 62 | 231
  Current smoker | 46 | 40 | 52 | 138
  Ex-smoker | 31 | 31 | 38 | 100
Alcohol Consumption [Number; unit: participants]
  Never | 49 | 54 | 51 | 154
  Once monthly or less often | 60 | 56 | 62 | 178
  Once per week | 26 | 20 | 21 | 67
  2 to 6 times per week | 24 | 22 | 14 | 60
  Daily | 1 | 5 | 4 | 10
Montgomery Åsberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression).
  scores on a scale | 33.4 (4.53) | 34.1 (4.07) | 33.7 (4.51) | 33.7 (4.37)
Hamilton Anxiety Scale Total Score [Mean (Standard Deviation); unit: scores on a scale] — Hamilton Anxiety Scale (HAM-A) is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (absent) to 56 (maximum severity).
  scores on a scale | 20.0 (6.14) | 20.1 (5.77) | 19.5 (5.42) | 19.9 (5.78)
Clinical Global Impression - Severity scale score [Mean (Standard Deviation); unit: sores on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  sores on a scale | 4.7 (0.61) | 4.7 (0.56) | 4.6 (0.59) | 4.7 (0.59)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a depression rating scale consisting of 10 items, each rated 0 (normal) to 6 (most abnormal). The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). A decrease in the total score or on individual items indicates improvement. Least squares (LS) means are from a mixed model for repeated measurements (MMRM) analysis of covariance (ANCOVA) with treatment, center, week, treatment-by-week interaction, Baseline MADRS total score-by-week as fixed effects.
Time Frame: Baseline and Week 8
Population: The full analysis set (FAS) included all randomized patients who received at least 1 dose of study drug, and had at least 1 valid post-baseline value for assessment of primary efficacy. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 15 mg
Number analyzed (Participants) | 126 | 123 | 113
scores on a scale | -12.87 (1.043) | -13.66 (1.064) | -13.36 (1.087)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; All statistical tests were 2-sided with the estimated P-values at the 5% level of significance. To control for multiplicity, a pre-specified sequential testing procedure for each dose was applied to compare 10 mg and 15 mg vortioxetine to placebo. Efficacy endpoints were tested for each dose in sequential order at significance level 0.025; as soon as an endpoint was non-significant at 0.025, the testing procedure stopped for all subsequent endpoints; Test type: Superiority or Other; p = 0.597, Mixed model for repeated measurements — Pre-specified sequential statistical testing procedure indicates that when p-value >0.025, hierarchical testing stops and for subsequent endpoints in the sequence a nominal p-value is provided; MMRM ANCOVA with treatment, center, week, treatment-by-week interaction, baseline MADRS total score-by-week as fixed effects; LS Mean Difference = -0.79, 95% CI 2-sided [-3.71 to 2.14], Standard Error of Mean 1.488
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 15 mg; Test type: Superiority or Other; p = 0.745, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.49, 95% CI 2-sided [-3.44 to 2.46], Standard Error of Mean 1.501

2. Secondary Outcome: Percentage of Participants With a MADRS Response at Week 8
Description: Response is defined as a participant with a ≥50% decrease in Montgomery Åsberg Depression Rating Scale (MADRS) total score from Baseline. The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). Decrease in the total score or on individual items indicates improvement.
Time Frame: Baseline and Week 8
Population: Full analysis set, last observation carried forward was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 15 mg
Number analyzed (Participants) | 149 | 143 | 142
percentage of participants | 32.9 | 37.8 | 37.3
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.396, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline MADRS score; Odds Ratio (OR) = 1.232, 95% CI 2-sided [0.761 to 1.995]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 15 mg; Test type: Superiority or Other; p = 0.435, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline MADRS score; Odds Ratio (OR) = 1.212, 95% CI 2-sided [0.748 to 1.963]

3. Secondary Outcome: Mean Clinical Global Impression Scale - Improvement (CGI-I) Score at Week 8
Description: The Clinical Global Impression - global improvement assesses the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. LS means were from a mixed model for repeated measurements (MMRM) ANCOVA with treatment, center, week, treatment-by-week interaction, Baseline Clinical Global Impression Scale-Severity of Illness (CGI-S) score-by-week as fixed effects.
Time Frame: Week 8
Population: The Full Analysis Set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 15 mg
Number analyzed (Participants) | 127 | 123 | 114
scores on a scale | 2.65 (0.105) | 2.56 (0.107) | 2.60 (0.110)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.554, Mixed model for repeated measurements; MMRM ANCOVA with treatment, center, week, treatment-by-week interaction, baseline CGI-S score-by-week as fixed effects; LS Mean Difference = -0.09, 95% CI 2-sided [-0.38 to 0.21], Standard Error of Mean 0.149
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 15 mg; Test type: Superiority or Other; p = 0.739, Mixed model for repeated measurements; MMRM ANCOVA with treatment, center, week, treatment-by-week interaction, baseline CGI-S score-by-week as fixed effects; LS Mean Difference = -0.05, 95% CI 2-sided [-0.35 to 0.25], Standard Error of Mean 0.151

4. Secondary Outcome: Change From Baseline in MADRS Total Score at Week 8 in Participants With Baseline Hamilton Anxiety Scale (HAM-A) Total Score ≥ 20
Description: The MADRS is a depression rating scale consisting of 10 items, each rated 0 (normal) to 6 (most abnormal). The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). A decrease in the total score or on individual items indicates improvement. LS means are from a mixed model for repeated measurements (MMRM) ANCOVA with treatment, center, week, treatment-by-week interaction, Baseline MADRS total score-by-week as fixed effects.
  HAM-A is a 14 item rating scale to quantify anxiety severity rated on a 5-point scale from 0 (not present) to 4 (severe) with a total score range from 0 to 56, where lower scores indicate mild severity.
Time Frame: Baseline and Week 8
Population: Full analysis set patients with a HAM-A Baseline score ≥ 20. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 15 mg
Number analyzed (Participants) | 60 | 57 | 56
scores on a scale | -14.11 (1.611) | -15.07 (1.650) | -12.37 (1.689)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.670, Mixed model for repeated measurements; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.97, 95% CI 2-sided [-5.43 to 3.50], Standard Error of Mean 2.261
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 15 mg; Test type: Superiority or Other; p = 0.451, Mixed model for repeated measurements; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.73, 95% CI 2-sided [-2.80 to 6.26], Standard Error of Mean 2.295

5. Secondary Outcome: Percentage of Participants in MADRS Remission at Week 8
Description: Remission is defined as a participant with a Montgomery Åsberg Depression Rating Scale (MADRS) total score ≤10. The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). Decrease in the total score or on individual items indicates improvement.
Time Frame: Week 8
Population: Full analysis set, last observation carried forward was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 15 mg
Number analyzed (Participants) | 149 | 143 | 142
percentage of participants | 22.1 | 26.6 | 23.9
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.352, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline MADRS total score; Odds Ratio (OR) = 1.291, 95% CI 2-sided [0.754 to 2.211]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 15 mg; Test type: Superiority or Other; p = 0.694, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline MADRS total score; Odds Ratio (OR) = 1.116, 95% CI 2-sided [0.646 to 1.928]

6. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score
Description: The Sheehan Disability Scale assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment. LS means were from mixed model for repeated measurements (MMRM) ANCOVA with treatment, center, week, treatment-by-week interaction, Baseline SDS total score-by-week as fixed effects.
Time Frame: Baseline and Week 8
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 15 mg
Number analyzed (Participants) | 77 | 74 | 62
scores on a scale | -9.38 (0.877) | -10.30 (0.959) | -8.69 (0.990)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.464, Mixed model for repeated measurements; MMRM ANCOVA with treatment, center, week, treatment-by-week interaction, baseline SDS total score-by-week as fixed effects; LS Mean Difference = -0.92, 95% CI 2-sided [-3.38 to 1.55], Standard Error of Mean 1.250
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 15 mg; Test type: Superiority or Other; p = 0.600, Mixed model for repeated measurements; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = 0.69, 95% CI 2-sided [-1.91 to 3.30], Standard Error of Mean 1.322

ADVERSE EVENTS:
Time Frame: A treatment-emergent adverse event is defined as any event whose onset occurs or intensity increases after the first dose of double-blind study medication through 30 days after permanent discontinuation of double-blind study medication.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 15 mg
Serious Adverse Events (participants affected / at risk) | 1/160 | 1/154 | 0/151
Other Adverse Events (participants affected / at risk) | 92/160 | 99/154 | 96/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=160) | Vortioxetine 10 mg (N=154) | Vortioxetine 15 mg (N=151)
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=160) | Vortioxetine 10 mg (N=154) | Vortioxetine 15 mg (N=151)
Vision blurred (Eye disorders) | 1 | 1 | 4
Nausea (Gastrointestinal disorders) | 17 | 47 | 51
Dry mouth (Gastrointestinal disorders) | 11 | 24 | 8
Vomiting (Gastrointestinal disorders) | 4 | 7 | 18
Constipation (Gastrointestinal disorders) | 6 | 16 | 14
Diarrhoea (Gastrointestinal disorders) | 10 | 10 | 15
Flatulence (Gastrointestinal disorders) | 4 | 10 | 5
Dyspepsia (Gastrointestinal disorders) | 5 | 3 | 3
Fatigue (General disorders) | 8 | 5 | 4
Irritability (General disorders) | 5 | 2 | 2
Pain (General disorders) | 4 | 1 | 1
Nasopharyngitis (Infections and infestations) | 8 | 6 | 3
Influenza (Infections and infestations) | 7 | 3 | 1
Viral upper respiratory tract infection (Infections and infestations) | 7 | 5 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 3
Bronchitis (Infections and infestations) | 4 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Headache (Nervous system disorders) | 29 | 24 | 25
Dizziness (Nervous system disorders) | 15 | 6 | 12
Tension headache (Nervous system disorders) | 3 | 7 | 3
Somnolence (Nervous system disorders) | 2 | 4 | 6
Insomnia (Psychiatric disorders) | 4 | 4 | 6
Anxiety (Psychiatric disorders) | 1 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4
Hot flush (Vascular disorders) | 6 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 6 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.